CLINICAL TRIAL: NCT03007368
Title: Assessment of Gastric Emptying and Fullness of Different Types of Foods in Mali
Brief Title: Digestion of Foods Consumed in Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1104010761
Record Dates: First submitted 2016-11-01; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Obesity and Other Hyperalimentation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Rice (Experimental): Cooked white rice and tomato-based sauce
  Interventions: Other: Rice
- Potato (Experimental): Cooked white peeled potato and tomato-based sauce
  Interventions: Other: Potato
- Pasta (Experimental): Cooked macaroni product and tomato-based sauce
  Interventions: Other: Pasta
- Sorghum thick porridge (Experimental): Sorghum thick porridge and tomato-based sauce
  Interventions: Other: Sorghum thick porridge
- Millet thick porridge (Experimental): Millet thick porridge and tomato-based sauce
  Interventions: Other: Millet thick porridge
- Millet couscous (Experimental): Cooked millet couscous and tomato-based sauce
  Interventions: Other: Millet couscous
- Millet thin porridge (Experimental): Millet thin porridge
  Interventions: Other: Millet thin porridge
- Millet thin monikuru porridge (Experimental): Millet thin porridge containing cooked millet granules (monikuru)
  Interventions: Other: Millet thin monikuru porridge

INTERVENTIONS:
Other: Rice — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Rice
Other: Potato — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response .
  Arms: Potato
Other: Pasta — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Pasta
Other: Sorghum thick porridge — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Sorghum thick porridge
Other: Millet thick porridge — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Millet thick porridge
Other: Millet couscous — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Millet couscous
Other: Millet thin porridge — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Millet thin porridge
Other: Millet thin monikuru porridge — Different modern and traditional starch-based foods found in Bamako, Mali were tested for differences in gastric emptying rate and appetitive response.
  Arms: Millet thin monikuru porridge

SUMMARY:
As populations become urbanized in Africa, the change to a more Westernized diet has been associated with rise in obesity and related metabolic syndrome diseases. The current study shows that in the West African Sahel, these replacement starchy staple foods have fast gastric emptying compared to traditional sorghum and millet foods; and implies that the latter could be beneficial in lowering glycemic response, providing energy from a meal over a longer time, and providing a satiety effect. Knowledge of this attribute of sorghum and millet foods could be useful to improve their image in West African cities to increase their consumption and to improve markets for local smallholder farmers.

DETAILED DESCRIPTION:
As suggested by anecdotal evidence that traditional Malian sorghum and millet foods are filling and provide sustained energy, we hypothesized that gastric emptying rates of sorghum and millet foods are slow, particularly compared to non-traditional starchy foods (white rice, potato, wheat pasta) that are now commonly consumed in urban areas of the West African Sahel. A broader purpose for the study was to understand whether sorghum and millet foods have positive health attributes that can be promoted in urban areas to provide better markets for local farmers.

Two human trials of similar design were conducted approximately one year apart. The carbon 13 (13C)-labelled octanoic acid breath test method was used to measure gastric emptying rate, and subjective pre-test and satiety response questionnaires were used. In the first study, 14 healthy volunteers in Bamako, Mali participated in a crossover design to test eight starchy foods for gastric emptying rate and satiety feelings. The second study with six volunteers was done to correct for endogenous 13C differences in the starch component of the foods.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (18 kg/m2 ≤ BMI ≤ 25 kg/m2)

Exclusion Criteria:

* Under any medication
* History of any gastrointestinal disease or surgery
* Diabetes
* Smoker

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Gastric emptying | acute study, 4 hours after consumption of test food
  Breath test was performed using 13C-octanoic acid mixed into test meals

SECONDARY OUTCOMES:
Appetitive response | acute study, 4 hours after consumption of test food
  Fullness and hunger questionnaire was given at various time points after consumption of test foods

IPD SHARING:
Plan to Share IPD: No
Not shared

REFERENCES:
- [Background] Ghoos YF, Maes BD, Geypens BJ, Mys G, Hiele MI, Rutgeerts PJ, Vantrappen G. Measurement of gastric emptying rate of solids by means of a carbon-labeled octanoic acid breath test. Gastroenterology. 1993 Jun;104(6):1640-7. doi: 10.1016/0016-5085(93)90640-x. PMID 8500721
- [Background] Choi MG, Camilleri M, Burton DD, Zinsmeister AR, Forstrom LA, Nair KS. [13C]octanoic acid breath test for gastric emptying of solids: accuracy, reproducibility, and comparison with scintigraphy. Gastroenterology. 1997 Apr;112(4):1155-62. doi: 10.1016/s0016-5085(97)70126-4. PMID 9097998
- [Background] Clegg ME, Shafat A. Procedures in the 13C octanoic acid breath test for measurement of gastric emptying: analysis using Bland-Altman methods. Scand J Gastroenterol. 2010 Aug;45(7-8):852-61. doi: 10.3109/00365521.2010.483740. PMID 20443742
- [Background] Schoeller DA, Klein PD, Watkins JB, Heim T, MacLean WC Jr. 13C abundances of nutrients and the effect of variations in 13C isotopic abundances of test meals formulated for 13CO2 breath tests. Am J Clin Nutr. 1980 Nov;33(11):2375-85. doi: 10.1093/ajcn/33.11.2375. PMID 6776794